CLINICAL TRIAL: NCT02296632
Title: Wireless Motion Sensors for Rheumatoid Arthritis Patients - Pilot Study and Preliminary Validation Effort
Brief Title: Wireless Motion Sensors for Rheumatoid Arthritis Patients - Pilot Study
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Brennan Spiegel, Director of Health Services Research, Cedars-Sinai Medical Center
Other Study IDs: Pro00036773
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Arthritis, Rheumatoid; Medication Adherence
Keywords: Telemedicine; Patient Reported Outcomes
MeSH Terms: conditions — Arthritis, Rheumatoid; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Motion sensors and daily online assessments — Patients will be asked to wear motion sensors during their waking hours and complete daily Patient Reported Outcomes online assessments.

SUMMARY:
This study aims to provide preliminary evidence of the validity of a sensor-based assessment of rheumatoid arthritis (RA) symptoms, and to collect structured qualitative feedback from RA Enbrel patients regarding the potential of a future biosensor/PRO mHealth application. The investigators' overarching hypothesis is that if patients have better and more timely information about whether Enbrel is working, then they will become more empowered and engaged in their treatment, more curious about how it may - or may not - be working, and potentially more compliant with therapy. However, this hypothesis remains largely untested.

DETAILED DESCRIPTION:
Patients with rheumatoid arthritis (RA) often endure a remitting and flaring disease-course characterized by considerable pain, stiffness, and fatigue. The social and emotional well-being of RA patients can suffer as a result. Data demonstrate that adherence to Enbrel significantly improves both functional status and health related quality of life (HRQOL) in RA patients. Yet patients prescribed Enbrel often exhibit non-adherence through early discontinuation, dose-stretching, and reduced persistence following medication "holidays". The knowledge, attitudes, and beliefs held by patients with regard to RA and Enbrel influence their perceptions of the benefits of, and barriers to, treatment.

Decisions to adhere occur when combined levels of susceptibility and severity provide the motivation to act, and the perception of benefits (less barriers) indicates a path of action. A given patient's ability to follow this path of action hinges on their relative self-efficacy: the conviction that they can successfully execute a behavior required to produce an expected outcome. Landscape literature reviews conducted by CORE-UCLA suggest that interventions targeting self-efficacy offer the greatest chance of improving adherence to Enbrel. Self-efficacy plays an important mediating role in self-management activities, allowing for the adoption and maintenance of health behaviors. Many studies have identified measures of self-efficacy as significant predictors of adherence in RA patients. Additionally - though with the caveat that they are methodologically heterogeneous and of limited generalizability - a number of studies have found that interventions targeting self-efficacy can significantly improve adherence related outcomes. Seminal works in the field - including Bandura's Social Cognition Theory and Rosenstock's Health Beliefs Model - have converged on the following recommendations for behavioral interventions targeting self-efficacy:

1. Identify and reinforce the patient's past and present successes or accomplishments.
2. Direct patients to observe successful behaviors and coping mechanisms of similar others, even if this involves having them alter or expand their social network.
3. Provide positive feedback for the patient's efforts or encourage people in the patient's social network, such as family members or friends, to do this.
4. Facilitate the patient in adopting new health behaviors by ensuring that patients do not interpret incorrectly how they are feeling.

Enabled by recent advances in microelectronics, signal processing algorithms, and networking capabilities, wireless health technologies hold the potential to support numerous aspects of these recommendations. Namely, motion sensors might contribute to the formation of a complete feedback loop involving self- monitoring, data presentation, and tailored messaging. Consumer Health Informatics (CHI) applications that offer complete feedback loops hold the most promise for improving self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Enbrel users between week -2 and week 5 of therapy, inclusive.
* Current active prescription for Enbrel with intent to use.
* 21 years or older.
* English speaking
* Have an understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

* Allergic to latex or dry natural rubber
* Using a pacemaker, implantable cardiac defibrillator, neurostimulator, hearing aids, cochlear implants or other electronic medical equipment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who are candidates to undergo treatment with the drug etanercept.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Qualitative measures of intervention experience | 28 days
  We will conduct in-person interviews with participants to learn about their experiences wearing motion sensors and completing daily online assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Spiegel, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Rosenstock, I. M. (1974). The health belief model and preventive health behavior. Health Education & Behavior, 2, 354-386.
- [Background] Bandura, A. (1996). Social foundations of thought and action: A social cognitive theory. Englewood Cliffs, NJ: Prentice Hall.
- [Background] Brus H, van de Laar M, Taal E, Rasker J, Wiegman O. Determinants of compliance with medication in patients with rheumatoid arthritis: the importance of self-efficacy expectations. Patient Educ Couns. 1999 Jan;36(1):57-64. doi: 10.1016/s0738-3991(98)00087-1. PMID 10036560
- [Background] Taal E, Rasker JJ, Seydel ER, Wiegman O. Health status, adherence with health recommendations, self-efficacy and social support in patients with rheumatoid arthritis. Patient Educ Couns. 1993 May;20(2-3):63-76. doi: 10.1016/0738-3991(93)90122-d. PMID 8337196
- [Background] Marks R, Allegrante JP, Lorig K. A review and synthesis of research evidence for self-efficacy-enhancing interventions for reducing chronic disability: implications for health education practice (part I). Health Promot Pract. 2005 Jan;6(1):37-43. doi: 10.1177/1524839904266790. PMID 15574526
- [Background] Rosenstock IM, Strecher VJ, Becker MH. Social learning theory and the Health Belief Model. Health Educ Q. 1988 Summer;15(2):175-83. doi: 10.1177/109019818801500203. PMID 3378902
- [Background] Gibbons MC, Wilson RF, Samal L, Lehman CU, Dickersin K, Lehmann HP, Aboumatar H, Finkelstein J, Shelton E, Sharma R, Bass EB. Impact of consumer health informatics applications. Evid Rep Technol Assess (Full Rep). 2009 Oct;(188):1-546. PMID 20629477
- [Background] Campbell, D. & Stanley, J. (1963). Experimental and quasi-experimental designs for research. Chicago, IL: Rand-McNally.
- [Background] Christodoulou C, Schneider S, Junghaenel DU, Broderick JE, Stone AA. Measuring daily fatigue using a brief scale adapted from the Patient-Reported Outcomes Measurement Information System (PROMIS (R)). Qual Life Res. 2014 May;23(4):1245-53. doi: 10.1007/s11136-013-0553-z. Epub 2013 Oct 17. PMID 24132347
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463